CLINICAL TRIAL: NCT07333391
Title: Evaluation of the Effectiveness of Individualized Grief Support Based on the Swanson Caring Model in Women Experiencing Pregnancy Loss
Brief Title: Individualized Grief Support With Swanson Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Fatma Pehlivan, Clinical Research Nurse, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SDUSuleyman
Record Dates: First submitted 2025-11-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Loss; Grief
Keywords: Pregnancy Loss; Grief; İndividualized care; Swanson model; Psychosocial Support

STUDY DESIGN:
Intervention Model Description: This research will be conducted as a mixed methods study involving both qualitative and quantitative methods. The qualitative part of the study will utilize a phenomenological design appropriate to the nature of the study, as part of a qualitative research design. The quantitative part of the study will be conducted as a randomized controlled trial. The sample consisted of 48 individuals who experienced pregnancy loss, agreed to participate in the study voluntarily, and met the inclusion criteria.Data will be collected using a Personal Information Form containing descriptive information about the women, the Perinatal Grief Scale (33-item short version), the Depression Anxiety Stress Scale-21 (DAS-21), and a semi-structured "Interview Form" based on the Swanson Model of Care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized and assigned to intervention and control groups based on the calculated number in the study.
  The Research Randomizer website was used to assign participants to the sample for determining the intervention and control groups. Research Randomizer is a free resource for researchers who need a quick way to generate random numbers or assign participants to experimental conditions (https://randomizer.org/).
  A sample randomization for a sample of 48 participants is as follows. Intervention Group 2, 3, 4, 5, 8, 10, 12, 13, 14, 15, 16, 20, 22, 25, 27, 29, 30, 34, 35, 40, 41, 43, 46, 47 Control Group
  1, 6,7, 9, 11, 17, 18, 19, 21, 23, 24, 26, 28, 31, 32, 33, 36, 37, 38, 39, 42, 44, 45, 48
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention: Control Group (No Intervention): Women assigned to the control group will be administered the Personal Information Form and pretests (PGS, DAS-21) at the first interview. Nurses will instruct the women on the hospital's routine procedures. No intervention will be administered. A posttest (PGS, DAS-21) will be administered three months after the loss.
- intervention group (Experimental): Women in the intervention group will complete a Personal Information Form and baseline measures (PGS, DAS-21) during the first hospital-based interview, where they will also receive an expert-informed grief brochure. One week after pregnancy loss, a second interview involving a semi-structured, phenomenological exploration of their grief experiences will be conducted. The 3rd, 4th, and 5th interviews-held three weeks after the second interview, in the second month, and in the third month-will focus on providing grief counseling and nursing care based on the Swanson care model. In the final interview, post-test measures (PGS, DAS-21) will be administered.
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Semi-structured interviews will be conducted with women who have experienced pregnancy loss, and their experiences and grieving processes will be examined phenomenologically. In the 3rd, 4th, and 5th interviews, based on the findings obtained from the qualitative data, grief counseling based on the Swanson care model will be provided to the women, and they will be provided with nursing care and grief support.
  Arms: intervention group

SUMMARY:
This study aims to examine the effects of individualized grief support for women experiencing pregnancy loss. The research, which will be conducted at Süleyman Demirel University, is a mixed-method design and includes both phenomenological qualitative analysis and randomized controlled quantitative trials. The sample will include 48 women; those with severe depression will be excluded. Quantitative data will be analyzed using SPSS, and qualitative data will be analyzed using content analysis.

DETAILED DESCRIPTION:
Pregnancy loss is a traumatic experience that leaves deep marks on women's lives. The grieving process that women experience during this period varies according to individual differences. The aim of this study is to examine the effects of individualized grief support for women who have experienced pregnancy loss. By addressing the emotional and psychological challenges women face after pregnancy loss, the study seeks to explore how the most appropriate support and care can be provided.

The sample of the study will consist of women who have experienced pregnancy loss at Süleyman Demirel University Research and Training Hospital, Department of Obstetrics and Gynecology. The power analysis of the study was conducted using the GPower 3.1.9.6 (Franz Faul, Universitaet Kiel, Germany) program, and the sample size was calculated as n=24+24=48. Women who obtain a very high score (14+) on the depression subscale of the Depression-Anxiety-Stress Scale will not be included in the study due to pathological findings.

This research will be conducted as a mixed-method study incorporating both qualitative and quantitative methods. In the qualitative part of the study, a phenomenological design, which is suitable for the nature of the research, will be used. The quantitative part will be conducted as a randomized controlled trial. Quantitative data are planned to be analyzed using the SPSS (Statistical Program for Social Sciences) 26.0 statistical analysis package. Qualitative data will be analyzed through content analysis using a software program commonly utilized for qualitative research.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above,
* Literate,
* Able to understand and speak Turkish,
* Desired and planned pregnancies
* No diagnosed psychiatric illness,
* No hearing or mental disabilit

Exclusion Criteria:

* Women who experienced pregnancy loss after infertility treatment
* Women who received psychological support during the process
* Women who scored very high on the DAS scale
* Women who withdrew from the study at any stage
* Women who did not complete the data collection forms will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who have experienced pregnancy loss
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form (Pre-Test) | At baseline (prior to intervention)
  This form will be administered to women during the initial interview after they are accepted into the service.
  It was developed by researchers to determine sociodemographic characteristics such as age, marital status, pregnancy history, and educational background. Women will also undergo pre-tests (PGS and DASS-21) during the initial interview.
Sociodemographic Characteristics Form | Baseline (pre-intervention)
  This form assesses participants' sociodemographic and obstetric characteristics, including age, marital status, educational level, and pregnancy history. The form is administered by the researcher during the initial interview after participants are accepted into the service.
Perinatal Grief Scale (PGS) Score | Baseline (pre-intervention)
  The Perinatal Grief Scale (PGS) is a self-report instrument used to assess grief intensity following pregnancy loss. The scale consists of 33 items rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 33 to 165, with higher scores indicating greater levels of perinatal grief.
Depression Anxiety Stress Scale-21 (DASS-21) | Baseline (pre-intervention)
  The Depression Anxiety Stress Scale-21 (DASS-21) is a self-report instrument used to assess symptoms of depression, anxiety, and stress. The scale consists of 21 items rated on a 4-point Likert scale ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The scale includes three subscales-Depression, Anxiety, and Stress-each comprising 7 items. Subscale scores are calculated by summing the relevant items and multiplying by two. Higher scores indicate greater symptom severity.
  Severity Classification:
  DASS-21 subscale scores are categorized as follows:
  Severity Level Depression Anxiety Stress Normal 0-4 0-3 0-7 Mild 5-6 4-5 8-9 Moderate 7-10 6-7 10-12 Severe 11-13 8-9 13-16 Extremely Severe ≥14 ≥10 ≥17
Bereavement Brochure | Immediately post-intervention
  A bereavement brochure, prepared with the contribution of experts, will be provided to women following pregnancy loss during the initial interview. The brochure contains information about emotional reactions, coping strategies, and available support resources.
Semi-Structured Interview | 1 week
  One week after the initial interview, semi-structured interviews will be conducted with women who have experienced pregnancy loss. In this interview, grief experiences and needs will be examined phenomenologically.
Swanson-Based Grief Counseling (First Session) | 3 weeks
  In the third interview, grief counseling will be provided based on findings from qualitative data. The counseling process will be structured using the Swanson Care Model.
Swanson-Based Bereavement Counseling (Second Session) | 2nd month
  In the fourth interview, bereavement counseling will again be conducted based on the Swanson Model, tailored to the woman's ongoing needs and responses.
Swanson-Based Bereavement Counseling (Third Session) + Post-Test Data Collection | 3rd month
  During the fifth interview, bereavement counseling will continue based on the Swanson Model. At this stage, post-test data collection forms (PGS and DASS-21) will also be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Taşçı Duran, Phd, RN, Study Director — Suleyman Demirel Üniversity
Locations (1):
- Suleyman Demirel University, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Bellhouse C, Temple-Smith MJ, Bilardi JE. "It's just one of those things people don't seem to talk about..." women's experiences of social support following miscarriage: a qualitative study. BMC Womens Health. 2018 Oct 29;18(1):176. doi: 10.1186/s12905-0 — https://pubmed.ncbi.nlm.nih.gov/30373583/
- See also: Hutti MH. Social and professional support needs of families after perinatal loss. J Obstet Gynecol Neonatal Nurs. 2005 Sep-Oct;34(5):630-8. doi: 10.1177/0884217505279998. PMID: 16227519. — https://pubmed.ncbi.nlm.nih.gov/16227519/
- See also: Koert E, Hartwig TS, Hviid Malling GM, Schmidt L, Nielsen HS. 'You're never pregnant in the same way again': prior early pregnancy loss influences need for health care and support in subsequent pregnancy. Hum Reprod Open. 2023 Aug 1;2023(3):hoad032. — https://pubmed.ncbi.nlm.nih.gov/37577178/
- See also: Lidegaard Ø, Mikkelsen AP, Egerup P, Kolte AM, Rasmussen SC, Nielsen HS. Pregnancy loss: A 40-year nationwide assessment. Acta Obstet Gynecol Scand. 2020 Nov;99(11):1492-1496. doi: 10.1111/aogs.13860. Epub 2020 Apr 26. PMID: 32255196. — https://pubmed.ncbi.nlm.nih.gov/32255196/
- See also: McSpedden M, Mullan B, Sharpe L, Breen LJ, Lobb EA. The presence and predictors of complicated grief symptoms in perinatally bereaved mothers from a bereavement support organization. Death Stud. 2017 Feb;41(2):112-117. doi: 10.1080/07481187.2016.1210696. — https://pubmed.ncbi.nlm.nih.gov/27573073/
- See also: Smith LK, Dickens J, Bender Atik R, Bevan C, Fisher J, Hinton L. Parents' experiences of care following the loss of a baby at the margins between miscarriage, stillbirth and neonatal death: a UK qualitative study. BJOG. 2020 Jun;127(7):868-874. — https://pubmed.ncbi.nlm.nih.gov/31976622/
- See also: Swanson KM. Effects of caring, measurement, and time on miscarriage impact and women's well-being. Nurs Res. 1999 Nov-Dec;48(6):288-98. doi: 10.1097/00006199-199911000-00004. PMID: 10571496. — https://pubmed.ncbi.nlm.nih.gov/10571496/
- See also: Zhuang S, Chen M, Ma X, Jiang J, Xiao G, Zhao Y, Hou J, Wang Y. The needs of women experiencing perinatal loss: A qualitative systematic review and meta-synthesis. Women Birth. 2023 Sep;36(5):409-420. doi: 10.1016/j.wombi.2023.03.007. Epub 2023 Apr 5. PM — https://pubmed.ncbi.nlm.nih.gov/37024379/
- See also: van den Berg MMJ, Dancet EAF, Erlikh T, van der Veen F, Goddijn M, Hajenius PJ. Patient-centered early pregnancy care: a systematic review of quantitative and qualitative studies on the perspectives of women and their partners. Hum Reprod Update. 2018 Ja — https://pubmed.ncbi.nlm.nih.gov/29040571/